CLINICAL TRIAL: NCT01612052
Title: Double Blinded Prospective Randomized Controlled Trial Comparing Cefazolin Plus Vancomycin Versus Cefazolin Plus Daptomycin for Vascular Surgery Prophylaxis
Brief Title: Vascular Surgical Antibiotic Prophylaxis Study (VSAPS 2)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Patrick Stone, MD, CAMC Medical Staff-with admitting privileges, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1997028
Record Dates: First submitted 2011-09-01; First posted 2012-06-05 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: MRSA - Methicillin Resistant Staphylococcus Aureus Infection
Keywords: Vascular Surgery
MeSH Terms: interventions — Antibiotic Prophylaxis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cefazolin plus Daptomycin (Active Comparator)
  Interventions: Drug: Antibiotic Prophylaxis
- Cefazolin plus Vancomycin (Active Comparator)
  Interventions: Drug: Antibiotic Prophylaxis

INTERVENTIONS:
Drug: Antibiotic Prophylaxis — Comparing the antibiotic treatment related to surgery

SUMMARY:
The current recommended antibiotic, Cefazolin, treatment for vascular surgery, provides coverage only for Methicillin-Sensitive Staphylococcus Aureaus (MSSA), other gram-positive bacteria, and some gram-negative bacteria which may not be adequate antibiotic treatment at the time of vascular surgery and result in an increased hospital length of stay, increased cost of care, and an increased risk of morbidity and mortality as a consequence of surgical site infections. Thus, the investigators want to compare whether Methicillin-resistant Staphylococcus Aureaus (MRSA) antibiotic prophylaxis with Cefazolin plus Daptomycin is superior to Cefazolin plus Vancomycin in the reduction of surgical site infection (SSI) following open arterial revascularization procedures requiring a groin plus lower extremity incision. The investigators hypothesis is that Cefazolin plus Daptomycin is superior to Cefazolin plus Vancomycin in the prevention of SSI for high risk patients undergoing open groin plus lower extremity procedures.

DETAILED DESCRIPTION:
There is an increase in surgical site infection (SSI) due to MRSA. The current recommended antibiotic, Cefazolin, treatment for vascular surgery, provides coverage only for Methicillin-Sensitive Staphylococcus Aureaus (MSSA), other gram-positive bacteria, and some gram-negative bacteria. To demonstrate that MRSA coverage is needed in vascular surgery with prosthetic graft placement in areas of the body that is at high risk for infection, the investigators are initiating a second study of patients undergoing groin plus lower extremity procedures by using combination antibiotics such as Cefazolin plus Daptomycin, Cefazolin plus Vancomycin. By decreasing post surgical site and prosthetic infections, the investigators could significantly reduce vascular surgery mortality and morbidity. Cost and amputation rates the investigators feel could also be reduced. Patients will be randomized in two groups -- Cefazolin plus Daptomycin, Cefazolin plus Vancomycin and will be evaluated during post procedure before discharge or within 30 days and between 30 and 360 days, for postoperative complications including cellulitis, graft infection, sepsis, limb loss, graft failure, and length of stay. If a patient is re-hospitalized, reason for the return and whether it is related to the procedure will be evaluated. Additionally, is there a graft failure, amputation, infection, hematoma, pseudoanurysm will be assessed. In case of a wound infection, the type of organism and finally, length of this hospitalization will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Any elective arterial revascularization procedure involving one or more groin plus lower extremity incisions
* Further, patient's considered at high risk because of history of MRSA colonization or infection, HIV, admission for >3 months in an acute care center or long-term care center will be included in the study.

Exclusion Criteria:

* Patient with an allergy to Cefazolin, Daptomycin or Vancomycin.
* Patients allergic to Penicillin.
* Patients enrolled in another IRB approved biomedical study.
* Patients with active infection requiring antibiotics preoperatively.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-03 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Difference between number of patients with MRSA infection between two groups | post procedure at 30 days

SECONDARY OUTCOMES:
Difference between number of patients with post-op complications between two groups | post procedure at 360 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stone, M.D., Principal Investigator — CAMC Medical Staff-with admitting privileges
Locations (1):
- Vascular Center of Excellence, Charleston, West Virginia, United States

REFERENCES:
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585